CLINICAL TRIAL: NCT02559778
Title: A Study Using Molecular Guided Therapy With Induction Chemotherapy Followed by a Randomized Controlled Trial of Standard Immunotherapy With or Without DFMO Followed by DFMO Maintenance for Subjects With Newly Diagnosed High-Risk Neuroblastoma
Brief Title: Pediatric Precision Laboratory Advanced Neuroblastoma Therapy
Acronym: PEDS-PLAN
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Giselle Sholler (Other)
Collaborators: Dell, Inc. (Industry); Beat NB Cancer Foundation (Other); K C Pharmaceuticals Inc. (Industry); Team Parker for Life (Unknown)
Responsible Party: Sponsor-Investigator, Giselle Sholler, Beat Childhood Cancer Chair, Milton S. Hershey Medical Center
Organization: Milton S. Hershey Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NMTRC012
Record Dates: First submitted 2015-09-22; First posted 2015-09-24 (Estimated); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — ceritinib; Dasatinib; Sorafenib; Vorinostat; Eflornithine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Immunotherapy without DFMO (Active Comparator): One of the following drugs will be chosen for each subject based on molecular guided results: ceritinib, dasatinib, sorafenib or vorinostat. This will be followed standard immunotherapy with Dinutuximab/GM-CSF/IL-2 and isotretinoin. At the end of immunotherapy, DFMO will be given to all subjects BID for 730 days.
  Interventions: Drug: Ceritinib; Drug: dasatinib; Drug: sorafenib; Drug: vorinostat
- Standard Immunotherapy with DFMO (Active Comparator): One of the following drugs will be chosen for each subject based on molecular guided results: ceritinib, dasatinib, sorafenib or vorinostat. This will be followed standard immunotherapy with Dinutuximab/GM-CSF/IL-2 and isotretinoin PLUS 1000mg/m2 BID of DFMO. At the end of immunotherapy, all subjects will go on to receive DFMO BID for 730 days.
  Interventions: Drug: Ceritinib; Drug: dasatinib; Drug: sorafenib; Drug: vorinostat; Drug: DFMO

INTERVENTIONS:
Drug: Ceritinib — One of the following drugs will be chosen for each subject based on molecular guided results: Ceritinib, dasatinib, sorafenib or vorinostat. This will be followed by consolidation, immunotherapy +/- DFMO, and then all subjects will receive DFMO for 2 years as maintenance.
  Other Names: Zykadia
Drug: dasatinib — One of the following drugs will be chosen for each subject based on molecular guided results: Ceritinib, dasatinib, sorafenib or vorinostat. This will be followed by consolidation, immunotherapy +/- DFMO, and then all subjects will receive DFMO for 2 years as maintenance.
  Other Names: Sprycel
Drug: sorafenib — One of the following drugs will be chosen for each subject based on molecular guided results: Ceritinib, dasatinib, sorafenib or vorinostat. This will be followed by consolidation, immunotherapy +/- DFMO, and then all subjects will receive DFMO for 2 years as maintenance.
  Other Names: Nexavar
Drug: vorinostat — One of the following drugs will be chosen for each subject based on molecular guided results: Ceritinib, dasatinib, sorafenib or vorinostat. This will be followed by consolidation, immunotherapy +/- DFMO, and then all subjects will receive DFMO for 2 years as maintenance.
  Other Names: ZOLINZA
Drug: DFMO — DFMO will be given to Arm B during immunotherapy and then for 2 years as maintenance to all subjects completing immunotherapy.
  Other Names: Eflornithine, α-difluoromethylornithine
  Arms: Standard Immunotherapy with DFMO

SUMMARY:
A prospective open label, multicenter study to evaluate the feasibility and acute toxicity of using molecularly guided therapy in combination with standard therapy followed by a Randomized Controlled Trial of standard immunotherapy with or without DFMO followed by DFMO maintenance for Subjects with Newly Diagnosed High-Risk Neuroblastoma.

ELIGIBILITY:
Part A- CLOSED:

1. Diagnosis: Subjects must have a diagnosis of neuroblastoma or ganglioneuroblastoma (nodular or intermixed) verified by histology or demonstration of clumps of tumor cells in bone marrow with elevated urinary catecholamine metabolites. Subjects with the following disease stages at diagnosis are eligible, if they meet the other specified criteria:

   a) Subjects with newly diagnosed neuroblastoma with INSS Stage 4 are eligible with the following: i. Age > 18 months (> 547 days) regardless of biologic features or ii. Age 12-18 months (365-547 days) with any of the following 3 unfavorable biologic features (MYCN amplification, unfavorable pathology and/or DNA index = 1) or iii. MYCN amplification (> 4-fold increase in MYCN signals as compared to reference signals), regardless of age or additional biologic features.

   b) Subjects with newly diagnosed neuroblastoma with INSS Stage 3 are eligible with the following: i. MYCN amplification (> 4-fold increase in MYCN signals as compared to reference signals), regardless of age or additional biologic features or ii. Age > 18 months (> 547 days) with unfavorable pathology, regardless of MYCN status.

   c) Subjects with newly diagnosed neuroblastoma with INSS Stage 2A/2B with MYCN amplification (> 4-fold increase in MYCN signals as compared to reference signals), regardless of age or additional biologic features.
2. Subjects must be age ≤ 21 years at initial diagnosis
3. Subjects must not have had prior systemic therapy except for localized emergency radiation to sites of life-threatening or function-threatening disease and/or no more than 1 cycle of chemotherapy per a low or intermediate risk neuroblastoma regimen (as per P9641, A3961, ANBL0531, or similar) prior to determination of MYCN amplification status and histology.
4. Specimens will be obtained only in a non-significant risk manner and not solely for the purpose of investigational testing.
5. Ability to tolerate PBSC collection: No known contraindication to PBSC collection. Examples of contraindications would include a weight or size less than that determined to be feasible at the collecting institution, or a physical condition that would limit the ability of the child to undergo apheresis catheter placement (if necessary) and/or the apheresis procedure.

   Part A and B both- Part A CLOSED, Part B- OPEN:
6. Adequate Cardiac Function Defined As:

   1. Shortening fraction of ≥ 27% by echocardiogram, or
   2. Ejection fraction of ≥ 50% by radionuclide evaluation or echocardiogram.
7. Adequate liver function must be demonstrated, defined as:

   c. Total bilirubin ≤ 1.5 x upper limit of normal (ULN) for age AND d. ALT (SGPT) < 10 x upper limit of normal (ULN) for age
8. Subjects must have adequate renal function defined as a serum creatinine based on age/gender as follows:

   Age Maximum Serum Creatinine (mg/dL) Male Female 1 month to < 6 months 0.4 0.4 6 months to < 1 year 0.5 0.5 1 to < 2 years 0.6 0.6 2 to < 6 year 0.8 0.8 6 to < 10 years 1 1 10 to < 13 years 1.2 1.2 13 to < 16 years 1.5 1.4

   ≥ 16 years 1.7 1.4
9. A negative serum pregnancy test is required for female participants of child bearing potential (≥13 years of age or after onset of menses)
10. Both male and female post-pubertal study subjects need to agree to use one of the more effective birth control methods during treatment and for six months after treatment is stopped. These methods include total abstinence (no sex), oral contraceptives ("the pill"), an intrauterine device (IUD), levonorgestrol implants (Norplant), or medroxyprogesterone acetate injections (Depo-provera shots). If one of these cannot be used, contraceptive foam with a condom is recommended.
11. Informed Consent: All subjects and/or legal guardians must sign informed written consent. Assent, when appropriate, will be obtained according to institutional guidelines.

    Part B- OPEN:
12. All patients must have a pathologically confirmed diagnosis of neuroblastoma, be age ≤ 21 years at initial diagnosis, and classified as high risk by the criteria used by COG or SIOPEN at the time of diagnosis. Exception: patients who are initially diagnosed as non-high-risk neuroblastoma, but later converted (and/or relapsed) to high risk neuroblastoma are also eligible.
13. Previous Therapy- subjects must fit into one of the strata categories listed in section 10.5 to be eligible to enroll on Part B of this study.
14. Pre-enrollment tumor survey:

    Prior to enrollment on Part B, a determination of mandatory disease staging must be performed. Tumor imaging studies including CT or MRI, MIBG or PET, and VMA/HVA (PET scan should be done for patients with prior disease that was MIBG non-avid). Bone marrow aspirates and biopsies are required.

    This disease assessment is required for eligibility and should be done preferably within 2 weeks, but must be done within a maximum of 4 weeks before first dose of study drug.
15. Timing- Enrollment to occur prior to Day + 120 post-transplant, preferably when the subject is within 28 days after completing local radiation therapy (if given).

Exclusion Criteria (Part A and B)

1. Subjects who are 12-18 months of age with INSS Stage 4 and all stage 3 subjects with favorable biologic features (ie, nonamplified MYCN, favorable pathology, and DNA index > 1) are not eligible.
2. Lactating females are not eligible unless they have agreed not to breastfeed their infants.
3. Subjects receiving any investigational drug concurrently.
4. Subjects with any other medical condition, including but not limited to malabsorption syndromes, mental illness or substance abuse, deemed by the Investigator to be likely to interfere with the interpretation of the results or which would interfere with a subject's ability to sign or the legal guardian's ability to sign the informed consent, and subject's ability to cooperate and participate in the study

Max Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 500 (Estimated)
Dates: Start 2015-09 (Actual); Primary Completion 2030-09 (Estimated); Study Completion 2035-09 (Estimated)

PRIMARY OUTCOMES:
Number of days from start of therapy to date of first relapse | Up to 8 years
  To measure the response of treatments chosen based on:
  • Event free survival (EFS)
Number of subjects that have a targeted agent chosen for treatment. | 2 years
  At completion of the induction therapy, the investigators will determine feasibility of adding molecularly guided targeted therapy to standard of care chemotherapy. Feasibility will be defined as:
  1. Subject has a targeted agent identified
  2. Receives 75% of dosing of medications while on study protocol during cycles 3-6
  3. Subject is not removed from study due to targeted agent drug related toxicity.
Number of subjects that receive 75% of dosing of medications while on study protocol during cycles 3-6. | 2 years
  At completion of the induction therapy, the investigators will determine feasibility of adding molecularly guided targeted therapy to standard of care chemotherapy. Feasibility will be defined as:
  1. Subject has a targeted agent identified
  2. Receives 75% of dosing of medications while on study protocol during cycles 3-6
  3. Subject is not removed from study due to targeted agent drug related toxicity.

SECONDARY OUTCOMES:
Number of days that subjects remain alive | 3 years plus 5 years follow up
  To measure the response of treatments chosen based on:
  * Overall response rate (ORR) after induction therapy
  * Overall survival (OS)
Overall Response Rate (ORR) of Participants by the presence of radiologically assessable disease by cross-sectional CT or MRI imaging and/or by MIBG or PET scans. | Up to 8 years
  To measure the response of treatments chosen based on:
  • Overall response rate (ORR) after induction therapy
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 3 years
  To compare toxicity effects of difluoromethylornithine (DFMO) in combination with Dinutuximab/GM-CSF/IL-2 and isotretinoin versus Dinutuximab/GM-CSF/IL-2 and isotretinoin alone.
Amount of pain medicine required by Arm A versus Arm B | 3 years
  To compare level of pain medicine needed during immunotherapy in patients receiving difluoromethylornithine (DFMO) in combination with Dinutuximab/GM-CSF/IL-2 and Isotretinoin versus those receiving Dinutuximab/GM-CSF/IL-2 and isotretinoin alone.
Number of subjects required to go off therapy due to treatment-related adverse events as assessed by CTCAE v4.0. | 1 year
  At completion of the induction therapy, the investigators will determine feasibility of adding molecularly guided targeted therapy to standard of care chemotherapy. Feasibility will be defined as:
  1. Subject has a targeted agent identified
  2. Receives 75% of dosing of medications while on study protocol during cycles 3-6
  3. Subject is not removed from study due to targeted agent drug related toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Giselle Sholler, MD, Study Chair — Beat Childhood Cancer
Locations (26):
- United States (25):
  - University of Alabama, Children's of Alabama, Birmingham, Alabama
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - UCSF Benioff Children's Hospital Oakland-, Oakland, California
  - Rady Children's Hospital, San Diego, California
  - Connecticut Children's Hospital, Hartford, Connecticut
  - Nicklaus Children's Miami, Miami, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - St. Joseph's Children's Hospital, Tampa, Florida
  - Augusta University Health, Augusta, Georgia
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - St. Lukes, Boise, Idaho
  - Advocate Children's Medical Group, Chicago, Illinois
  - University of Louisville, Louisville, Kentucky
  - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Children's Hospital and Clinics of Minnesota, Minneapolis, Minnesota
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Levine Children's Hospital, Charlotte, North Carolina
  - Randall Children's Hospital, Portland, Oregon
  - Penn State Milton S. Hershey Medical Center and Children's Hospital, Hershey, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Dell Children's Blood and Cancer Center, Austin, Texas
  - Children's Medical Center, Dallas, Texas
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
- UHC Sainte-Justine, Montreal, Quebec, Canada

REFERENCES:
- See also: Beat Childhood Cancer Main Website — http://beatcc.org